CLINICAL TRIAL: NCT00606515
Title: A Clinical Trial to Compare the Pharmacokinetics of Two Formulations of Taxane, Paclitaxel Injection and Liposomal Paclitaxel, in Humans
Brief Title: Pharmacokinetics Study of Liposomal Paclitaxel in Humans
Acronym: LPS-PK-H
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Luye Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Dr. Li Jin, Cancer Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: LPS-PK-01-2008
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Cancer
Keywords: Pharmacokinetics; Liposomal paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Liposomal paclitaxel
  Interventions: Drug: Liposomal paclitaxel
- B (Active Comparator): Paclitaxel
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Liposomal paclitaxel — Patients will be given Liposomal paclitaxel intravenously in 3 hours with the dose of 175mg/m2 at the first day of chemotherapy. Cycle duration will be 21 days. Each patient will receive 3 cycles of therapy.
  Arms: A
Drug: Paclitaxel — Patients will be given paclitaxel intravenously in 3 hours with the dose of 175mg/m2 at the first day of chemotherapy. Cycle duration will be 21 days. Each patient will receive 3 cycles of therapy.
  Arms: B

SUMMARY:
The purpose of this study is to determine whether there is any difference of the pharmacokinetics of two taxane formulations, paclitaxel injection and liposomal paclitaxel in Chinese cancer patients with solid tumors.

DETAILED DESCRIPTION:
The pharmacokinetics of a new formulation of taxane (liposomal paclitaxel) has never been studied in Chinese cancer patients. This clinical trial is designed to find out the pharmacokinetics of liposomal paclitaxel at the dose of 175mg/m2 and whether it has a different pharmacokinetic profile to paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have histologically confirmed solid tumors of advanced stages
* Patients who are suitable for being treated with liposomal paclitaxel only
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Patients who are expected to be alive for at least 3 months
* Adequate hematologic, hepatic and renal functions
* Adequate other organ functions as defined by the protocol
* No prior systemic chemotherapy at least 4 weeks before the recruitment
* No previous anaphylactic reaction to hormone.

Exclusion Criteria:

* Allergy to any study medication
* Serious complication that would compromise the patient's ability to complete the study
* Grade ≥1 neuropathy using NCI CTCAE version 3.0 criteria
* Pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 72 hours after the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Doctor, Principal Investigator — Cancer Hospital of Fudan University
Locations (2):
- China (2):
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Cancer Hospital of Fudan University, Shanghai